CLINICAL TRIAL: NCT01616433
Title: Arthritis Foundation Exercise Program & "10 Keys" to Healthy Aging
Brief Title: Arthritis Foundation Exercise Program & "10 Keys" to Healthy Aging--Prevention Research Center
Acronym: AFEP+10 Keys
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IU48DP09-0014918-01
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Arthritis; Diabetes; Hypertension; Preventive Behaviors
Keywords: Arthritis; Preventive Behaviors
MeSH Terms: conditions — Arthritis; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arthritis Foundation Exercise Program (Active Comparator)
  Interventions: Behavioral: AFEP
- AFEP + 10 Keys to Healthy Aging (Experimental): Arthritis Foundation Exercise Program integrated with the "10 Keys" to Healthy Aging
  Interventions: Behavioral: "10 Keys" to Healthy Aging

INTERVENTIONS:
Behavioral: AFEP — Arthritis Foundation Exercise Program (10 weeks, twice a week, 60 minutes per session)
  Other Names: Arthritis Foundation Exercise Program (10 weeks, twice a week, 60 minutes per session)
  Arms: Arthritis Foundation Exercise Program
Behavioral: "10 Keys" to Healthy Aging — "10 Keys" to Healthy Aging. 10 week program, twice a week, 75 minutes per session.
  Arms: AFEP + 10 Keys to Healthy Aging

SUMMARY:
Older adults are at high risk for loss of independence because of age-related chronic health conditions. Of these chronic conditions, arthritis accounts for the largest proportion of the disability in the community. The investigators propose to target older adults who have self-reported arthritis or joint pain for dissemination of a disability prevention program. The program will be a collaborative effort of the Arthritis Foundation, the investigators Prevention Research Center staff and other key partners in the community. The project will develop information needed to provide guidance for implementation of the investigators intervention by other agencies and organizations. As a major thrust of the investigators CDC Prevention Research Center, the investigators have developed a comprehensive program focused on preventing disease and disability in older adults: the "10 Keys to Healthy Aging". Each of the 10 Keys disseminates proven approaches and current recommendations for prevention in older adults, focusing on age 65+ but also addressing age 50-65 years. The overall objective is to determine if an integrated evidence based exercise intervention (AFEP) combined with health education on preventive practices for older adults ("10 Keys") is more effective for improving mobility and risk factors for mobility disability and use of preventive services compared to exercise alone (AFEP). The investigators will also propose to evaluate the impact of geographic location on outcomes and overall sustainability of the program.

ELIGIBILITY:
Inclusion Criteria:

* 50+ years old
* Attends at last one exercise class in a 10 week program

Exclusion Criteria:

* On oxygen
* Hospitalized for cardiac event in past 6 months (at least 1 overnight)
* Had major surgery in past 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Preventive Behaviors | 1 year
  Measuring preventive behaviors emphasized by the "10 Keys" to Healthy Aging, such as cancer screenings, controlling blood pressure, immunizations, etc.
Joint Pain & Stiffness | 1 year
  Self-reported joint pain and stiffness, as measured by the WOMAC.
Cholesterol (LDL) | 1 year
  LDL cholesterol
Glucose | 1 year
  Fasting glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Community sites, Allegheny County Primarily, Pennsylvania, United States